CLINICAL TRIAL: NCT03548558
Title: Testing Means to Scale Early Childhood Development Interventions in Rural Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Lunenfeld Tanenbaum Research Institute (Other); Safe Water and AIDS Project (Other); University of California, Berkeley (Other); McGill University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jill Luoto, Research Scientist, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01HD090045 (NIH); R21HD098508 (NIH); R01HD090045 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-06-07 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Early Child Development
Keywords: Early Childhood Development; Parenting Behaviors; Group-based curriculum; Kenya; Child Outcomes; Community Health Volunteers

STUDY DESIGN:
Intervention Model Description: The evaluation design is conducted in two phases. During phase 1, a clustered Randomized Control Trial (cRCT) across 60 community health volunteers (CHVs) and their associated villages are randomly assigned to one of three equally-sized treatment arms: group meetings for 16 biweekly sessions over 8 months (Arm 1), 12 group meetings plus 4 home visits over 8 months (Arm 2), and a control group (Arm 3). Within half of villages assigned to Arms 1 and 2, fathers will also be invited to the sessions (a 2x2 factorial design among the 40 villages assigned to receive the intervention). After a first follow-up survey immediately after the end of the biweekly sessions, in phase 2 we stratify by Arms 1 and 2 and re-randomize villages so that 20 total receive booster group sessions every 2 months over another 2 years (10 each from Arms 1 and 2). The other 20 villages from Arms 1 and 2 do not receive extended boosters.
Who Masked: Outcomes Assessor
Masking Description: The study will have separate teams for collection of surveys and program implementation. Due to the nature of the intervention, the participants and delivery agents will not be blinded to their study allocation as part of the program implementation team. Data collectors of surveys for the research team will, however, be blinded to the intervention allocation status of participants and villages. (Baseline surveys will be collected prior to randomization.) Likewise, data analysis will be blinded to the intervention status of participants and villages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Arm 1 ("group" sessions) (Experimental): Group meetings only (16 total)
  Interventions: Behavioral: Group sessions
- Arm 2 ("group+home" sessions) (Experimental): Mixed group meetings with a limited number of individual home visits (12 group meetings + 4 home visits)
  Interventions: Behavioral: Group+Home sessions
- Arm 3 (No Intervention): This arm will serve as the control group to identify the effects of a parenting intervention and the most effective mode of delivery, as well as the sustained impacts from the intervention
- Arm B (Booster villages) (Experimental): In one half of Arm 1 and Arm 2 villages above, after the end of the main intensive intervention, extended light-touch group booster sessions held every other month over two years between the two follow-up surveys will be held
  Interventions: Behavioral: Group sessions; Behavioral: Group+Home sessions; Behavioral: Booster sessions
- Arm A (Non-booster villages) (Other): In the other half of Arm 1 and Arm 2 villages, no boosters will be held during phase 2
  Interventions: Behavioral: Group sessions; Behavioral: Group+Home sessions
- Arm X: Fathers invited (Experimental): During phase 1, fathers were invited to attend sessions in half of Arms 1 and 2 villages.
  Interventions: Behavioral: Group sessions; Behavioral: Group+Home sessions; Behavioral: Fathers invited
- Arm Y: Fathers not invited (Other): During phase 1, fathers were not invited in the other half of Arms 1 and 2 villages.
  Interventions: Behavioral: Group sessions; Behavioral: Group+Home sessions

INTERVENTIONS:
Behavioral: Group sessions — Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 8 months. CHVs will record attendance at each session. To maximize participation, prior to each session the CHVs will send a short message service (SMS) mobile phone reminder of the session's topic, time and location to all participants.
  Arms: Arm 1 ("group" sessions); Arm A (Non-booster villages); Arm B (Booster villages); Arm X: Fathers invited; Arm Y: Fathers not invited
Behavioral: Group+Home sessions — Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV.
  Arms: Arm 2 ("group+home" sessions); Arm A (Non-booster villages); Arm B (Booster villages); Arm X: Fathers invited; Arm Y: Fathers not invited
Behavioral: Booster sessions — After the end of the 16 biweekly sessions (phase 1), we will re-randomize across the 40 intervention villages, stratified by Arms 1 and 2, and half of each of Arm 1 and Arm 2 villages will receive group booster visits every other month for the period between end-line and follow-up surveys. This will constitute Phase 2 of the study.
  Arms: Arm B (Booster villages)
Behavioral: Fathers invited — During phase 1's 16 biweekly sessions, in half of Arm 1 and Arm 2 villages (20 total), fathers will additionally be invited to attend the 16 sessions. Separate father-only sessions will be held for 4 of the 16 sessions. This randomization will end after phase 1.
  Arms: Arm X: Fathers invited

SUMMARY:
This study aims to experimentally test the effectiveness and cost-effectiveness of competing models of delivery of an Early Childhood Development (ECD) intervention in rural Kenya to determine how to maximize their reach to improve child cognitive, language and relevant psychosocial outcomes. The study will also include a longer-term evaluation of sustained impacts; an examination of the pathways of change leading to intervention impacts to inform policy; and examination of the role of paternal involvement on child development. Findings will provide policy makers with rigorous evidence of how best to expand ECD interventions in low-resource rural settings to improve child developmental outcomes for both the short-and longer-term.

DETAILED DESCRIPTION:
Recent neurobiological and psychological research has established that vital development occurs in language, cognitive, motor and socio-emotional development during the first few years of life, and early life outcomes are key determinants of adult outcomes such as educational achievement, labor market outcomes, and health. Yet more than 200 million children under age five in low and middle income countries (LMICs) will fail to reach their developmental potential as adults, predominantly due to poverty, poor health and nutrition, and inadequate cognitive and psychosocial stimulation. Early childhood development (ECD) interventions that integrate nutrition and child stimulation activities have been proposed as a powerful policy tool for the remediation of early disadvantages in poor settings, and numerous field studies have shown they can be effective in improving children's developmental and health outcomes, at least in the short-term. Key questions remain on what models of delivery are the most effective and cost-effective that can be potentially scalable in LMICs, as well as how to sustain parental behavioral changes over time, which can lead to long-term improvements in child development and the possibility of positive spillovers to benefit younger siblings. Having a better understanding of the underlying behavioral pathways leading from intervention, to parental behavior changes, to child impacts, is also key to inform policy about the optimal design of interventions to maximize their scalability and sustainability. This study will conduct a multi-arm clustered randomized controlled trial across 60 villages and 1200 households in rural Western Kenya that tests different potentially cost-effective delivery models for an ECD intervention with a curriculum that integrates child psychosocial stimulation and nutrition education. Selected households will undergo baseline and follow-up surveys to measure short-term impacts in parental behaviors and children's developmental outcomes, and the study will collect data on potential mediators of parental behavioral change to uncover the pathways leading to impacts. Two follow-up surveys, one immediately after the end of the planned intervention and a second two years later, will enable testing of the short term and midterm sustainability of impacts, as well as the presence of any spillovers onto younger siblings. In collaboration with a local non-governmental organization (NGO), the Safe Water and AIDS Project (SWAP), community health volunteers (CHVs) will be trained to implement the intervention by introducing the ECD curriculum in their villages.

The goal of this study is to provide policymakers with rigorous evidence of how best to expand ECD interventions in low-resource rural settings.

ELIGIBILITY:
Inclusion Criteria:

* Kenyan mothers or equivalent female primary caretakers aged 15 and over with children aged 6-24 months (classified as mature minors)
* Kenyan fathers aged 18 and older with children aged 6-24 months with a mother present

The unit of observation for the study is the household or family, within which the primary focus is mother-child dyads and household eligibility hinges on the age of the child. For those households with a father present, the study will additionally include him in some analyses and surveys.

Exclusion Criteria:

* Households without children
* Households with children that are outside the age range of 6-24 months at baseline
* Households with a mother younger than 15 or one aged 15-18 still living with her parents
* Single fathers

Selection criteria for fathers are based on the mother-child eligibility criteria. Fathers will be included if and when appropriate per the details surrounding the mother-child dyads.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill E. Luoto, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC, Los Angeles, California, United States

REFERENCES:
- [Derived] Lopez Garcia I, Saya UY, Luoto JE. Cost-effectiveness and economic returns of group-based parenting interventions to promote early childhood development: Results from a randomized controlled trial in rural Kenya. PLoS Med. 2021 Sep 28;18(9):e1003746. doi: 10.1371/journal.pmed.1003746. eCollection 2021 Sep. PMID 34582449
- [Derived] Luoto JE, Lopez Garcia I, Aboud FE, Singla DR, Zhu R, Otieno R, Alu E. An Implementation Evaluation of A Group-Based Parenting Intervention to Promote Early Childhood Development in Rural Kenya. Front Public Health. 2021 May 5;9:653106. doi: 10.3389/fpubh.2021.653106. eCollection 2021. PMID 34026713
- [Derived] Luoto JE, Lopez Garcia I, Aboud FE, Singla DR, Fernald LCH, Pitchik HO, Saya UY, Otieno R, Alu E. Group-based parenting interventions to promote child development in rural Kenya: a multi-arm, cluster-randomised community effectiveness trial. Lancet Glob Health. 2021 Mar;9(3):e309-e319. doi: 10.1016/S2214-109X(20)30469-1. Epub 2020 Dec 17. PMID 33341153
- [Derived] Luoto JE, Lopez Garcia I, Aboud FE, Fernald LCH, Singla DR. Testing means to scale early childhood development interventions in rural Kenya: the Msingi Bora cluster randomized controlled trial study design and protocol. BMC Public Health. 2019 Mar 4;19(1):259. doi: 10.1186/s12889-019-6584-9. PMID 30832624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1265 households assessed for eligibility during a household census exercise immediately preceding baseline survey (60 village clusters across 3 sub-counties)
Pre-assignment Details: Of 1265 assessed for eligibility, 1152 households were enrolled into the study and randomized to an intervention arm in phase 1. This included 1152 mothers, 1152 children, and 512 fathers at baseline. Analysis performed at level of households. Excluded households included 52 who migrated away, 20 refusals, 6 children had a physical or mental impairment and 35 households were unavailable after 3 visit attempts. Between phase 1 and 2, father arm washed out and replaced with booster randomization.
Units Other Than Participants: Cluster RCT at Village Level Assignment
Groups:
- Arm 1 "Groups" Without Fathers: Group meetings only (16 total) for phase 1. Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 8 months for Phase 1. Fathers are not invited (10 total villages).
- Arm 1 "Groups" With Fathers: 10 total villages had group sessions and invited fathers during Phase 1's 16 biweekly sessions
- Arm 2 ("Group+Home" Sessions) Without Fathers: Mixed group meetings with a limited number of individual home visits (12 group meetings + 4 home visits)
  Group+Home sessions: During phase 1, households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Fathers not invited. 10 villages total.
- Arm 2 "Group + Home" Sessions, With Fathers Invited: Mixed group meetings with a limited number of individual home visits (12 group meetings + 4 home visits)
  Group+Home sessions: During phase 1, households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Fathers will also be invited. 10 villages total.
- Arm B (Booster Villages) (Phase 2): In one half of Arm 1 and Arm 2 villages above, after the end of the main intensive intervention, extended light-touch group booster sessions held every other month over two years between the two follow-up surveys will be held during phase 2.
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 7 months. CHVs will record attendance at each session. To maximize participation, prior to each session the CHVs will send a short message service (SMS) mobile phone reminder of the session's topic, time and location to all participants.
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV.
- Arm A (Non-booster Villages) Phase 2: In the other half of Arm 1 and Arm 2 villages, no boosters will be held
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 7 months. CHVs will record attendance at each session. To maximize participation, prior to each session the CHVs will send a short message service (SMS) mobile phone reminder of the session's topic, time and location to all participants.
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV.
Period: Phase 1: 16 Total Fortnightly Sessions
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Started | 173; 10 Cluster RCT at Village Level Assignment (173 households with 173 mothers, 173 children, and 70 fathers enrolled at baseline.) | 202; 10 Cluster RCT at Village Level Assignment (202 households with 202 mothers, 202 children, and 90 fathers enrolled at baseline.) | 201; 10 Cluster RCT at Village Level Assignment (201 households with 201 mothers, 201 children, and 87 fathers enrolled at baseline.) | 199; 10 Cluster RCT at Village Level Assignment (199 households with 199 mothers, 199 children, and 103 fathers enrolled at baseline.) | 377; 20 Cluster RCT at Village Level Assignment (377 households with 377 mothers, 377 children, and 162 fathers enrolled at baseline.) | 0; 0 Cluster RCT at Village Level Assignment (Booster village assignments were randomized after first phase to begin phase 2. Half of arm 1 and arm 2 villages were re-randomized into receiving boosters at this stage for a total of 20 villages, half from each of Arms 1 and 2.) | 0; 0 Cluster RCT at Village Level Assignment (Booster village assignments were randomized after first phase to begin phase 2. Half of arm 1 and arm 2 villages were re-randomized into receiving boosters at this stage for a total of 20 villages, the other 20 villages did not receive supplemental boosters.)
Completed | 161; 10 Cluster RCT at Village Level Assignment | 185; 10 Cluster RCT at Village Level Assignment | 191; 10 Cluster RCT at Village Level Assignment | 182; 10 Cluster RCT at Village Level Assignment | 351; 20 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment
Not Completed | 12; 0 Cluster RCT at Village Level Assignment | 17; 0 Cluster RCT at Village Level Assignment | 10; 0 Cluster RCT at Village Level Assignment | 17; 0 Cluster RCT at Village Level Assignment | 26; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment
Not completed — Death | 2 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 7 | 15 | 9 | 13 | 24 | 0 | 0
Period: Phase 2: Booster Sessions Every 2 Months
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Started | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 377; 20 Cluster RCT at Village Level Assignment (All originally enrolled households assigned to control villages remained eligible for inclusion in phase 2) | 394; 20 Cluster RCT at Village Level Assignment (All originally enrolled households at baseline remained eligible for phase 2. Boosters were re-randomized across Arms 1 and 2 at conclusion of phase 1. The starting sample size of 394 for this phase subtracts 3 deaths that occurred between baseline and the first follow-up survey in these villages. Fathers not enrolled for phase 2.) | 378; 20 Cluster RCT at Village Level Assignment (All originally enrolled households at baseline remained eligible for phase 2. Boosters were re-randomized across Arms 1 and 2 at conclusion of phase 1. The starting sample size for this phase subtracts 1 death that occurred between baseline and the first follow-up survey in these villages. Fathers not enrolled for phase 2.)
Completed | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 308; 20 Cluster RCT at Village Level Assignment | 323; 20 Cluster RCT at Village Level Assignment (There was 1 additional death between follow-up surveys 1 and 2 for booster villages.) | 313; 20 Cluster RCT at Village Level Assignment (There was 1 additional death between follow-up survey waves in non-booster villages.)
Not Completed | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 0; 0 Cluster RCT at Village Level Assignment | 69; 0 Cluster RCT at Village Level Assignment | 71; 0 Cluster RCT at Village Level Assignment | 65; 0 Cluster RCT at Village Level Assignment
Not completed — Death | 0 | 0 | 0 | 0 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 62 | 67 | 61

BASELINE CHARACTERISTICS:
Population: Booster randomization came after baseline in a 2x2 design with the original randomization to one of the 3 main study arms. 1152 refers to number of households (mother-child dyads) enrolled into study.
Groups:
- Arm 1 ("Group" Sessions) Without Fathers: Group meetings only (16 total)
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 8 months. Fathers not invited.
- Arm 1 ("Group" Sessions) With Fathers: Group meetings only (16 total)
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 8 months. Fathers will be invited.
- Arm 2 ("Group+Home" Sessions) Without Fathers: Mixed group meetings with a limited number of individual home visits (12 group meetings + 4 home visits)
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV. Fathers not invited.
- Arm 2 ("Group+Home" Sessions) With Fathers: Mixed group meetings with a limited number of individual home visits (12 group meetings + 4 home visits) plus fathers invited.
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV. Fathers invited.
- Arm B (Booster Villages): In one half of Arm 1 and Arm 2 villages above, after the end of the main intensive intervention, extended light-touch group booster sessions held every other month over two years between the two follow-up surveys will be held during phase 2.
- Total: Total of all reporting groups
Arm/Group | Arm 1 ("Group" Sessions) Without Fathers | Arm 1 ("Group" Sessions) With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 ("Group+Home" Sessions) With Fathers | Arm 3 | Arm B (Booster Villages) | Arm A (Non-booster Villages) | Total
Number analyzed (Participants) | 173 | 202 | 201 | 199 | 377 | 0 | 0 | 1152
Age, Continuous [Mean (Standard Deviation); unit: Months] — Child age at baseline in months
  Months | 13.5 (5.2) | 14.1 (4.8) | 14.3 (4.7) | 14.6 (4.7) | 14.2 (4.7) |  |  | 14.2 (4.8)
Age, Customized [Mean (Standard Deviation); unit: years] — Maternal age in years. Father's age was not systematically recorded.
  years
    Maternal age in years | 28.7 (9.0) | 28.0 (9.1) | 28.7 (8.9) | 27.7 (7.6) | 29.2 (9.0) |  |  | 28.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex breakdown for the children targeted by intervention at baseline. All children were enrolled alongside their mothers or other female primary caretaker. A total of 512 fathers were enrolled at baseline as well, all males. Population: Recruitment and eligibility for study participation centered on mothers with eligible children. A total of 512 fathers were surveyed at baseline alongside mothers and children out of 1152 mother-child dyads originally recruited into the study. Numbers analyzed for fathers therefore lower.
  Participants
    Child Sex: Female | 82 | 95 | 96 | 92 | 185 |  |  | 550
    Child Sex: Male | 91 | 107 | 105 | 107 | 192 |  |  | 602
    Mother Sex: Female | 173 | 202 | 201 | 199 | 377 |  |  | 1152
    Mother Sex: Male | 0 | 0 | 0 | 0 | 0 |  |  | 0
    Father sex (baseline): number analyzed (Participants) | 70 | 90 | 87 | 103 | 162 | 0 | 0 | 512
    Father sex (baseline): Female | 0 | 0 | 0 | 0 | 0 |  |  | 0
    Father sex (baseline): Male | 70 | 90 | 87 | 103 | 162 |  |  | 512
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/ethnicity information for the targeted and enrolled child at baseline, mothers, and enrolled fathers at baseline. Numbers of participants at household level analyzed.
  Participants
    Black : Children | 173 | 202 | 201 | 199 | 377 |  |  | 1152
    Black : Mothers | 173 | 202 | 201 | 199 | 377 |  |  | 1152
    Black : Fathers | 70 | 90 | 87 | 103 | 162 |  |  | 512
Region of Enrollment [Number; unit: Households/enrolled children] — Recorded at level of targeted/enrolled child (household level).
  Households/enrolled children
    Kenya | 173 | 202 | 201 | 199 | 377 |  |  | 1152
Child cognitive score (Bayley III) [Mean (Standard Deviation); unit: units on a scale (0-19)] — The Bayley Scales of Infant Development 3rd edition (Bayley's III), is validated in African settings and provides measures for all dimensions of child development up to 42 months of age. The official age-standardized cognitive and receptive language scales have 0-19 range with higher values denoting better scores.
  units on a scale (0-19)
    Baseline age-standardized cognitive scores | 9.0 (2.3) | 9.6 (2.1) | 9.2 (2.2) | 9.8 (2.3) | 9.5 (2.3) |  |  | 9.4 (2.2)
    Baseline age-standardized receptive language scores | 9.2 (2.1) | 9.4 (2.3) | 9.2 (1.8) | 10.0 (2.4) | 9.7 (2.3) |  |  | 9.5 (2.2)
Family Care Indicators (FCI) [Median (Standard Deviation); unit: score on a scale] — At baseline, the study will use the Family Care Indicators, a self-reported measure of parenting practices which measures the quality time spent with children in learning and playing activities for young children at home. Scores range 0-12. Higher values are considered to be better.
  score on a scale | 4.8 (2.2) | 4.7 (2.0) | 4.4 (1.9) | 4.8 (2.0) | 5.0 (2.0) |  |  | 4.8 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Child Developmental Outcomes
Description: The Bayley Scales of Infant Development 3rd edition (Bayley's III), is validated in African settings and provides measures for all dimensions of child development up to 42 months of age. The official age-standardized cognitive, receptive language, and expressive language scales have 0-19 ranges with higher values denoting better scores. At month 11/endline survey, cognitive, receptive language, and expressive language scales were collected. At baseline, cognitive and receptive language were collected. Month 11 reported here. Baseline outcomes reported elsewhere.
Time Frame: Month 11/Endline after end of Phase 1's 16 biweekly sessions (Arm 1 with & without fathers, Arm 2 with and without fathers, and Arm 3). Arms A and B created after the Month 11/Endline survey.
Population: Arms A and B created after the Month 11/Endline survey after re-randomizing among Arms 1 and 2 (with and without fathers)
Measure: Mean (Standard Deviation); unit: age-standardized scores on a scale
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Number analyzed (Participants) | 161 | 185 | 191 | 182 | 351 | 0 | 0
age-standardized scores on a scale
  Age-standardized cognitive score at month 11/endline survey | 9.5 (1.8) | 9.4 (1.7) | 9.1 (1.5) | 9.1 (1.6) | 8.7 (1.5) |  |
  Age-standardized receptive language score at month 11/endline survey | 10.6 (2.3) | 10.5 (2.2) | 10.0 (1.7) | 10.2 (1.9) | 9.7 (1.8) |  |
  Age-standardized expressive language score at month 11/endline survey | 8.8 (138) | 9.0 (1.6) | 8.6 (1.7) | 8.6 (1.5) | 8.9 (1.7) |  |

2. Primary Outcome: Child Developmental Outcomes
Description: Block-design subtest of the Wechsler Preschool and Primary Scale of Intelligence - 4th Edition (WPPSI-IV) to measure cognitive non-verbal reasoning. This subtest produces an age-standardized scaled score that can range from 1 to 19, with higher scores denoting better outcomes. For expressive and receptive language we used Dholuo and Kiswahili versions of the British Picture Vocabulary Scale - III (BPVS III), which includes 168 items for use with ages 3-17 years old. Knowledge of receptive vocabulary is measured by asking the respondent to point to one of four pictures that corresponds to a word (object, person, or action) spoken by the assessor; for expressive vocabulary the assessor pointed to a picture and the child named it. Pictures were adapted to the Kenyan context previously. Raw language scale ranges 0-25 with higher values denoting better outcomes.
Time Frame: Month 35-37/Follow-Up survey (Arms 3, A and B), two years after end of Phase 1's 16 biweekly sessions
Population: Analyzed those children who were successfully tracked until this Month 35-37 survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 308 | 323 | 313
scores on a scale
  Block Design WPPSI-III |  |  |  |  | 4.9 (2.1) | 5.2 (2.2) | 5.1 (2.1)
  BPVS receptive language |  |  |  |  | 14.4 (4.2) | 14.5 (4.2) | 14.4 (4.3)
  BPVS expressive language |  |  |  |  | 10.5 (3.2) | 10.4 (2.9) | 10.6 (3.1)

3. Primary Outcome: Parenting Practices (HOME Observation for Measurement of the Environment - HOME)
Description: At follow-up surveys, the study will collect the Home Observation for Measurement of the Environment (HOME)- Short Form (SF) inventory. The HOME-SF includes items grouped into two sub-scales: emotional support and cognitive stimulation. It has four parts: one for children under age three; a second for children between the ages of three and five; a third for children ages six through nine; and a fourth version for children ten and over. The total raw score for the HOME-SF is a simple summation of the recorded individual item scores and it varies by age group, as the number of individual items varies according to the age of the child. At the endline/month 11 survey the HOME scale scores ranged from 0-45, with higher scores denoting better outcomes.
Time Frame: Month 11/Endline survey (Arm 1 with and without fathers, Arm 2 with and without Fathers, Arm 3).
Population: Sample sizes at month 11/endline survey. Arms A and B created after this survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Number analyzed (Participants) | 161 | 185 | 191 | 182 | 351 | 0 | 0
score on a scale | 30.2 (5.6) | 31.6 (5.9) | 32.4 (5.2) | 30.9 (6.1) | 28.9 (6.2) |  |

4. Primary Outcome: Parenting Practices (HOME Observation for Measurement of the Environment - HOME)
Description: At follow-up surveys, the study will collect the Home Observation for Measurement of the Environment (HOME)- Short Form (SF) inventory. The HOME-SF includes items grouped into two sub-scales: emotional support and cognitive stimulation. It has four parts: one for children under age three; a second for children between the ages of three and five; a third for children ages six through nine; and a fourth version for children ten and over. The total raw score for the HOME-SF is a simple summation of the recorded individual item scores and it varies by age group, as the number of individual items varies according to the age of the child. At the month 35-37/follow-up survey the HOME score ranged 0-55 with higher scores denoting better outcomes.
Time Frame: Month 35-37 Follow-up Survey (Arms 3, A and B).
Population: Sample sizes at month 35-37/follow-up survey two years after end of Phase 1's 16 biweekly sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 308 | 323 | 313
score on a scale |  |  |  |  | 36.7 (6.9) | 38.5 (6.4) | 37.6 (6.5)

5. Secondary Outcome: Child Height
Description: child length-for-age measured in centimeters. Enumerators measured the child three times and calculated the mean; all measures were converted to length-for-age Z scores following World Health Organization (WHO) recommendations and calculated using Stata version 16's "zscore06" command that uses 2006 WHO child growth standards and adjusts for child age and sex. Mean score is 0 for reference population. A score of <-2 SD is considered stunted linear growth. Higher scores represent better outcomes.
Time Frame: Month 11/endline survey.
Population: At month 11/endline survey, child length-for-age was measured for a total of 1053 children out of 1070.
Measure: Mean (Standard Deviation); unit: z-score length-for-age
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Number analyzed (Participants) | 159 | 182 | 190 | 180 | 342 | 0 | 0
z-score length-for-age | -1.39 (1.09) | -1.42 (1.00) | -1.43 (1.04) | -1.46 (1.14) | -1.29 (1.08) |  |

6. Secondary Outcome: Changes in Nutritional Practices
Description: Child dietary diversity is measured using a 0-7 scale in which parents report the categories of foods eaten by the child in the past 24 hours following WHO recommendations for child feeding. Higher scores denote better dietary diversity.
Time Frame: Month 11/endline survey (Arms 1, 2 with and without fathers, and Arm 3), and follow-up 2/month 35-37 survey (Arms 3, A and B).
Population: Dietary diversity data collected for 1063 mother-child dyads at month 11/endline survey, and 942 dyads at two-year follow-up/month 35-37 survey. Arms A and B only analyzed at month 35-37 survey, Arms 1 & 2 only at month 11/endline survey.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 "Groups" Without Fathers | Arm 1 "Groups" With Fathers | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 "Group + Home" Sessions, With Fathers Invited | Arm 3 | Arm B (Booster Villages) (Phase 2) | Arm A (Non-booster Villages) Phase 2
Number analyzed (Participants) | 161 | 184 | 190 | 181 | 347 | 323 | 313
scores on a scale
  Dietary diversity at month 11/endline survey: number analyzed (Participants) | 161 | 184 | 190 | 181 | 347 | 0 | 0
  Dietary diversity at month 11/endline survey | 4.3 (1.1) | 4.3 (1.2) | 4.1 (1.1) | 4.0 (1.1) | 4.1 (1.2) |  |
  Dietary diversity at follow-up 2/month 35-37 survey: number analyzed (Participants) | 0 | 0 | 0 | 0 | 306 | 323 | 313
  Dietary diversity at follow-up 2/month 35-37 survey |  |  |  |  | 3.8 (1.1) | 3.7 (1.3) | 3.7 (1.3)

7. Other Pre Specified Outcome: Changes in Perceived Social Support
Description: The study will measure perceived social support using the Duke-University of North Carolina (UNC) Functional Social Support Questionnaire, which is a multidimensional, self-administered instrument that assesses the social support that a person perceives that he or she has. The social support is measured as 2 scales for confidant or affective support.
Time Frame: Baseline, 10-12, and 22-24 months after intervention
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Relationship Support Scale
Description: a 10-item measure self-reported by the mother on relationship quality with her husband using a 3-point scale from "rarely" to "most days" experiencing things ranging from the husband insulting the wife to the husband helping with child care.
Time Frame: Baseline, 10-12, and 22-24 months after intervention
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in Problem Solving/Social Support
Description: Daily stress will be assessed using the Daily Stress Index which measures on a 0-2 scale (never, sometimes, often) the difficult things that sometimes happen to people. This index has previously been used in Uganda, and the raw score will be aggregated over the 15 parts with a range of 0-30.
Time Frame: Baseline, 10-12, and 22-24 months after intervention
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Maternal Depression
Description: The study will measure maternal psychological well-being using the widely used Center for Epidemiologic Studies Depression Scale (CESD) with proven psychometric properties. The 20-item scale examines how individuals have felt in the previous week. The options include: 0= Rarely (0-1 days); 1= Some or a little of the time (at least 1-2 days); 2= Most of the days (3 or more days). Scoring is done as follows: zero for answers in the first option, 1 for answers in the second option, 2 for answers in the third option. The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Time Frame: Baseline, 10-12, and 22-24 months after intervention
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Maternal Knowledge
Description: The study will elicit maternal knowledge about child development through asking mothers about the ages at which they think the child would be able achieve certain developmental milestones, which are then compared with the expected ages reported in the literature.
Time Frame: Baseline, 10-12, and 22-24 months after intervention
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in Maternal Beliefs
Description: The study will adapt and measure the scale to elicit beliefs developed by Cunha et al. (2013)with the target of eliciting parental beliefs regarding the benefits of providing children better cognitive and non-cognitive stimulation. The instrument asks parents about developmental milestones in language and socio-emotional development under different home scenarios, which are constructed using data from the Family Care Indicators.
Time Frame: Baseline, 10-12, and 22-24 months after intervention
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Changes in Self-efficacy
Description: The Self-Efficacy for Parenting Tasks Index-Toddler Scale (SEPTI-TS) is a 26-item questionnaire to assess parental self-efficacy in parents of toddlers. The Short Form of the SEPTI-TS showed a strong factor structure with four subscales of domain-specific parental self-efficacy (Nurturance, Discipline, Play, and Routine) that showed high reliability. Scores are rates from strongly disagree to strongly agree, and higher scores indicate stronger parental self-efficacy
Time Frame: Baseline, 10-12, and 22-24 months after intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Arms 1 and 2, with and without fathers, up to 13 months, then up to 2 years after re-randomization of Arms 1 and 2 into Arms A and B. Adverse Events were collected from Arm 3 throughout the entire study period, up to 37 months.
Groups:
- Arm 1 ("Group" Sessions) Without Fathers Invited: Group meetings only (16 total)
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 8 months. 10 villages total. Fathers not invited.
- Arm 1 ("Group" Sessions) With Fathers Invited: Group meetings only (16 total)
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 8 months. 10 villages total. Fathers also invited.
- Arm 2 ("Group+Home" Sessions) Without Fathers: Mixed group meetings with a limited number of individual home visits (12 group meetings + 4 home visits)
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV. 10 villages total, fathers not invited.
- Arm 2 ("Group + Home" Sessions) With Fathers Invited: Mixed group meetings with a limited number of individual home visits (12 group meetings + 4 home visits)
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV. 10 villages total, fathers also invited.
- Arm B (Booster Villages): In one half of Arm 1 and Arm 2 villages above, after the end of the main intensive intervention, extended light-touch group booster sessions held every other month over two years between the two follow-up surveys will be held
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 7 months. CHVs will record attendance at each session. To maximize participation, prior to each session the CHVs will send a short message service (SMS) mobile phone reminder of the session's topic, time and location to all participants.
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV.
- Arm A (Non-booster Villages): In the other half of Arm 1 and Arm 2 villages, no boosters will be held
  Group sessions: Mother-child dyads in Arm 1 households will receive biweekly ECD sessions for a total of 16 sessions over 7 months. CHVs will record attendance at each session. To maximize participation, prior to each session the CHVs will send a short message service (SMS) mobile phone reminder of the session's topic, time and location to all participants.
  Group+Home sessions: Households in Arm 2 will receive a total of 16 sessions with identical content similar to Arm 1, but 4 of those sessions will replace group sessions held at the level of villages for personalized home visits, in which the CHV will visit each participant household to deliver these sessions. These home visits will cover identical material and topics as the group sessions in Arm 1 villages, but will be delivered on a personalized basis in the home of the mother and child. Personal barriers to the practices will be discussed and an active resolution strategy developed in concert with the CHV.
Arm/Group | Arm 1 ("Group" Sessions) Without Fathers Invited | Arm 1 ("Group" Sessions) With Fathers Invited | Arm 2 ("Group+Home" Sessions) Without Fathers | Arm 2 ("Group + Home" Sessions) With Fathers Invited | Arm 3 | Arm B (Booster Villages) | Arm A (Non-booster Villages)
All-Cause Mortality (participants affected / at risk) | 2/173 | 1/202 | 0/201 | 1/199 | 3/377 | 1/394 | 1/378
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/202 | 0/201 | 0/199 | 0/377 | 0/394 | 0/378
Other Adverse Events (participants affected / at risk) | 0/173 | 0/202 | 0/201 | 0/199 | 0/377 | 0/394 | 0/378

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT03548558/Prot_SAP_000.pdf